CLINICAL TRIAL: NCT05428592
Title: A Randomized, Blinded, Parallel-controlled Phase 3 Study to Evaluate the Immunogenicity and Safety of SARS-CoV-2 mRNA Vaccine (LVRNA009) as Heterologous Booster in Participants Aged 18 Years and Older Vaccinated 2 Doses Inactivated SARS-CoV-2 Vaccine
Brief Title: Clinical Trial of SARS-CoV-2 mRNA Vaccine(LVRNA009) as Heterologous Booster in Islamabad
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AIM Vaccine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LVRNA009-Ⅲ-02
Record Dates: First submitted 2022-06-14; First posted 2022-06-23 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — LVRNA009 COVID-19 vaccine; sinovac COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: A randomized, blinded, parallel-controlled design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVRNA009 study group (Experimental)
  Interventions: Biological: LVRNA009
- CoronaVac® control group (Active Comparator)
  Interventions: Biological: CoronaVac®

INTERVENTIONS:
Biological: LVRNA009 — 50μg /0.5 mL/Vial/person
  Arms: LVRNA009 study group
Biological: CoronaVac® — 0.5 mL/Vial, 0.5mL per human dose containing 600SU of inactivated SARS-CoV-2 antigen
  Arms: CoronaVac® control group

SUMMARY:
This study is a randomized, blinded, parallel-controlled phase 3 clinical trial. The study intent to evaluate the immunogenicity and safety of SARS-CoV-2 mRNA Vaccine (LVRNA009) as heterologous booster in participants aged 18 years and older vaccinated 2 doses Inactivated SARS-CoV-2 Vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older.
2. Understand the contents of the ICF and voluntarily sign it (If the participant is unable to sign the ICF on his/her own due to illiteracy, an impartial witness is needed).
3. Participants who are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, and other study procedures.
4. Female participants of childbearing potential or partners of male participants: voluntarily agree to use effective contraception with their partners 14 days prior to the vaccination and must agree to continue such precautions during the study until 3 months after vaccination. [Effective contraception includes oral contraceptives, injectable or implantable contraception, extended-release topical contraceptives, hormonal patches, intrauterine devices (IUDs), sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.].
5. For female participants: without childbearing potential (amenorrhea for at least 1 year or documented surgical sterilization) or have used effective contraception with a negative pregnancy test before vaccination in this study.
6. Axillary temperature <37.3°C/99.1°F at screening visit and 72 hours prior to vaccination.
7. Healthy participants or participants with mild underlying disease [in a stable state without exacerbation (no admission to hospital or no major adjustment to treatment regimen, etc.) for at least 3 months prior to enrollment in this study].
8. Participants who have vaccinated 2 doses of CoronaVac® (with an interval of 3-8 weeks between 2 doses), for 6-12 months prior to enrollment.

Exclusion Criteria:

1. Previous medications intervention for the prophylaxis or prevention of COVID-19 (Including vaccination with any licensed SARS-CoV-2 vaccines other than 2 doses of CoronaVac® ).
2. History of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS) or other coronavirus infections.
3. History of a previous laboratory-confirmed diagnosis of SARS-CoV-2 infection or COVID-19.
4. History of allergy to any component of the study vaccine or history of severe allergic reaction to the vaccine or drug (including but not limited to anaphylaxis, allergic laryngeal oedema, anaphylactic purpura, thrombocytopenic purpura, or localized allergic necrosis (Arthus reaction)).
5. Positive nucleic acid for SARS-CoV-2 in nasopharyngeal/oropharyngeal swab specimens.
6. Positive HIV test result.
7. A history or family history of convulsions, epilepsy, encephalopathy and psychosis.
8. Malignant tumors in the active phase, malignant tumors not receiving adequate treatment, malignant tumors at potential risk of recurrence during the study period.
9. Congenital or functional splenic deficiency, complete or partial splenectomy for any reason.
10. Prolonged (defined as more than 14 days) use of immunosuppressive or other immunomodulatory drugs (e.g., corticosteroids, ≥20 mg/d prednisone or equivalent; however, inhaled and topical steroids are permitted) within 6 months prior to the vaccine.
11. Any other licensed vaccines given within 28 days prior to the study vaccination, or planned administration of vaccine(s) within 28 days after vaccination.
12. Have received immunoglobulin or other blood products within 3 months prior to enrollment or plan to receive them during the study period.
13. Blood donation or blood loss ≥ 450 mL within 1 month prior to enrolment, or planned donation during the study period.
14. Participants who have received any other investigational product within 1 month prior to enrollment or intent to participate in another clinical study at any time during the conduct of this study.
15. Female participants who are pregnant or breastfeeding.
16. Participants deemed unsuitable for participation in this study based on the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 (Wild-type strain) VNA (live virus neutralizing assay) | 14 days after vaccination for all participants
Seroconversion Rate (SCR) of SARS-CoV-2 (Wild-type strain) VNA (live virus neutralizing assay) | 14 days after vaccination for all participants
  Seroconversion is defined as: GMT post vaccination≥ 4-fold rise from baseline GMT value
Incidence of each solicited (local and systemic) AE and each unsolicited AE | AE within 14 days, unsolicited AE within 28 days after vaccination for all participants
Intensity of each solicited (local and systemic) AE and each unsolicited AE | AE within 14 days, unsolicited AE within 28 days after vaccination for all participants
Duration of each solicited (local and systemic) AE and each unsolicited AE | AE within 14 days, unsolicited AE within 28 days after vaccination for all participants

SECONDARY OUTCOMES:
Geometric mean increase (GMI) of SARS-CoV-2 (Wild-type strain) VNA (live virus neutralizing assay) | 14 days after vaccination for all participants
GMT of SARS-CoV-2 (Wild-type strain) VNA (live virus neutralizing assay) | 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
SCR of SARS-CoV-2 (Wild-type strain) VNA (live virus neutralizing assay) | 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
GMI of SARS-CoV-2 (Wild-type strain) VNA (live virus neutralizing assay) | 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
GMT of SARS-CoV-2 (Wild-type strain) VNA (pseudo-virus neutralizing assay) | 14 days, 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
SCR of SARS-CoV-2 (Wild-type strain) VNA (pseudo-virus neutralizing assay) | 14 days, 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
GMI of SARS-CoV-2 (Wild-type strain) VNA (pseudo-virus neutralizing assay) | 14 days, 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
GMT of S-protein specific IgG antibodies (ELISA) | 14 days, 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
SCR of S-protein specific IgG antibodies (ELISA) | 14 days, 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
GMI of S-protein specific IgG antibodies (ELISA) | 14 days, 28 days, 3 months, 6 months, and 12 months after vaccination for all participants
Incidence of serious adverse events (SAEs), adverse events of special interest (AESI), and the occurrence of pregnancy events | within 12 months after vaccination for all participants
Intensity of serious adverse events (SAEs), adverse events of special interest (AESI), and the occurrence of pregnancy events | within 12 months after vaccination for all participants
Causality of serious adverse events (SAEs), adverse events of special interest (AESI), and the occurrence of pregnancy events | within 12 months after vaccination for all participants

OTHER OUTCOMES:
Cellular immune subgroup: virus antigen-specific IL-2, IL-4, IL-13, IFN-γ cytokine titers (ELISpot) | 7 days, 14 days, and 28 days after vaccination
Cross-neutralization subgroup: cross-neutralizing ability of VNA (live virus neutralizing assay) against other VOCs of SARS-CoV-2 | 14 and 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Aamer Ikram, Principal Investigator — National Institute of Health, Islamabad
Locations (1):
- Clinical Trial Unit, National Institute of Health, Islamabad, Pakistan